CLINICAL TRIAL: NCT05382728
Title: A Phase III, Randomised, Double-blind, Multi-center Study to Assess the Efficacy and Safety of TY-9591 Tablets Versus Osimertinib as First Line Treatment in Patients With EGFR-sensitive Mutation, Locally Advanced or Metastatic Non Small Cell Lung Cancer.
Brief Title: Phase III Study of TY-9591 in Patients With Locally Advanced or Metastatic Non-small Cell Lung Cancer (FLETEO)
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: TYK Medicines, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TYKM1601301
Record Dates: First submitted 2022-05-16; First posted 2022-05-19 (Actual); Last update posted 2024-01-30 (Actual); Status verified 2024-01

CONDITIONS: NSCLC; EGFR Activating Mutation
MeSH Terms: interventions — osimertinib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TY-9591+placebo Osimertinib (Experimental): TY-9591 (160mg orally, once daily) plus placebo Osimertinib (80mg orally, once daily), in accordance with the randomization schedule.
  Interventions: Drug: TY-9591; Drug: placebo Osimertinib
- Osimertinib+placebo TY-9591 (Active Comparator): Osimertinib (80mg orally, once daily) plus placebo TY-9591 (160mg orally, once daily), in accordance with the randomization schedule.
  Interventions: Drug: Osimertinib; Drug: placebo TY-9591

INTERVENTIONS:
Drug: TY-9591 — The dose of TY-9591 is 160 mg once daily. A cycle of treatment is defined as 21 days of once daily treatment.
  Number of Cycles: as long as patients are continuing to show clinical benefit, as judged by the Investigator, and in the absence of discontinuation criteria.
  Other Names: TY-9591 Tablets
  Arms: TY-9591+placebo Osimertinib
Drug: placebo Osimertinib — The dose of placebo Osimertinib is 80 mg once daily. A cycle of treatment is defined as 21 days of once daily treatment.
  Number of Cycles: as long as patients are continuing to show clinical benefit, as judged by the Investigator, and in the absence of discontinuation criteria.
  Other Names: placebo Tagrisso
  Arms: TY-9591+placebo Osimertinib
Drug: Osimertinib — The dose of Osimertinib is 80 mg once daily. A cycle of treatment is defined as 21 days of once daily treatment.
  Number of Cycles: as long as patients are continuing to show clinical benefit, as judged by the Investigator, and in the absence of discontinuation criteria.
  Other Names: Tagrisso
  Arms: Osimertinib+placebo TY-9591
Drug: placebo TY-9591 — The dose of placebo TY-9591 is 160 mg once daily. A cycle of treatment is defined as 21 days of once daily treatment.
  Number of Cycles: as long as patients are continuing to show clinical benefit, as judged by the Investigator, and in the absence of discontinuation criteria.
  Other Names: placebo TY-9591 Tablets
  Arms: Osimertinib+placebo TY-9591

SUMMARY:
To assess the efficacy and safety of TY-9591 versus Osimertinib in patients with locally advanced or Metastatic Non Small Cell Lung Cancer.

DETAILED DESCRIPTION:
This is a Phase III, double-blind, randomised study assessing the efficacy and safety of TY-9591 versus Osimertinib in patients with locally advanced or metastatic Non-small Cell Lung Cancer (NSCLC) that is known to be EGFR sensitising mutation (EGFRm) positive, treatment-naïve and eligible for first-line treatment with an EGFR-TKI.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female aged ≥18 years and <80 years.
2. Locally advanced or metastatic NSCLC diagnosed by histology or cytology.
3. Presence of an activating EGFR-sensitive mutations (including exon 19 deletions, L858R, the above mentioned mutations alone or co-existed with other EGFR-mutated sites).
4. No prior systemic antitumor therapy for locally advanced or metastatic NSCLC.
5. At least one measurable lesion according to Response Evaluation Criteria in Solid Tumours (RECIST) version 1.1.
6. The ECOG score is 0-1, and there is no deterioration 2 weeks before the study, and the expected survival is not less than 3 months.
7. Adequate bone marrow reserve function, and no liver, kidney and coagulation dysfunction.
8. Male patients and female patients of reproductive age should take adequate contraceptive measures from signing informed consent to 3 months after the last study drug treatment; Women of childbearing age have negative pregnancy test results within 7 days of the first dose.
9. Patients having recovered from all grade ≤ 1 toxicities related to previous anticancer therapies (CTCAE v 5.0) except for alopecia, platinum-therapy-related neuropathy (where ≤2 is allowed) before first dose of study treatment.
10. Patients can understand and voluntarily sign the informed consent form.
11. Patient able to comply with study requirements.

Exclusion Criteria:

1. Any of the following treatment:

   1. Previous treatment with EGFR inhibitor;
   2. Previous treatment with Systematic antitumor therapy (including targeted therapy, biotherapy and immunodrug therapy, etc.)；
   3. Previous treatment with standard chemotherapy with 28 days before the first dose of the study drug, and traditional Chinese medicine antitumor therapy within 7 days before the first dose of the study drug;
   4. Receiving radiation to more than 30% of the bone marrow or with a wide field of radiation that had to be completed within 28 days of the first dose of study treatment; Radiotherapy with a limited field of radiation within 7 days of the first dose of study treatment or palliative radiation therapy for bone metastasis;
   5. Uncontrollable or poorly controlled pleural and abdominal effusion;
   6. Major surgery within 28 days of the first dose of study treatment;
   7. Patients currently receiving (or at least within 14 days prior to receiving the first dose )medications or herbal supplements known to be potent inhibitors or inducers of cytochrome P450 isoenzyme (CYP)3A4;
   8. Patients who are receiving and need to continue receiving medications during the study that are known to prolong the QTc interval or may cause tachycardia;
   9. Participants in other clinical trials (other than non-interventional clinical trials) within 28 days prior to the first administration of the investigational drug.
2. Pathologically confirmed squamous cell carcinoma or squamous cell component predominance in NSCLC.
3. Symptomatic brain metastases or leptomeningeal metastases.
4. Patients have spinal cord compression caused by tumor.
5. Clinically severe gastrointestinal dysfunction may affect the ingestion, transport or absorption of the study drugs.
6. Cardiac function and disease are consistent with the following:

   1. Corrected QT interval(QTc)≥ 470 milliseconds from 3 times of electrocardiograms (ECGs);
   2. Any clinically important abnormalities in rhythm;
   3. Any factors that increase the risk of QTc prolongation;
   4. Left ventricular ejection fraction (LVEF) <50%.
7. Active human immunodeficiency virus (HIV), syphilis, hepatitis c virus (HCV) or hepatitis b virus (HBV) infection, with the exception of asymptomatic chronic hepatitis b or hepatitis c carriers.
8. Previous history of interstitial lung disease(ILD), drug-induced ILD or radiation pneumonitis require steroid treatment, or any evidence of clinically active ILD diseases.
9. Previous allogeneic bone marrow transplant.
10. Pregnant or lactating women.
11. Any other disease or medical condition that is unstable or may affect the safety or study compliance.
12. Hypersensitivity to investigational drug or similar compounds or excipients.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 680 (Estimated)
Dates: Start 2022-06-08 (Actual); Primary Completion 2025-05 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Median Progression Free Survival (PFS) | approximately 18 months
  PFS is defined as time from randomization until the date of first documented disease progression or death due to any cause

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | approximately 18 months
  ORR is defined as the proportion of patients with a best overall response of complete response (CR) or partial response (PR) during the study treatment
Intracranial Overall Response Rate (iORR) | approximately 18 months
  iORR is defined as the proportion of patients with a best intracranial response of complete response (CR) or partial response (PR) during the study treatment
Intracranial Median Progression Free Survival (iPFS) | approximately 18 months
  iPFS is defined as time from randomization until the date of first documented intracranial disease progression or death due to any cause
Duration of Response (DoR) | approximately 18 months
  DoR is defined as the time from the date of first documented response (PR or CR) until the date of first documented disease progression or death due to any cause during the study treatment
Disease Control Rate (DCR) | approximately 18 months
  DCR is defined as the proportion of patients with a best overall response of complete response (CR) , partial response (PR) or Stable disease (SD) ≥6 weeks during the study treatment
Clinical Benefit Rate (CBR) | approximately 18 months
  CBR is defined as the proportion of patients with a best overall response of complete response (CR) , partial response (PR) or Stable disease (SD) ≥24 weeks during the study treatment
Depth of Response (DepOR) | approximately 18 months
  The Depth of response was defined as the relative change in the sum of the longest diameters of Response Evaluation Criteria in Solid Tumors (RECIST) Target lesions (TLs) at the nadir compared to baseline, in the absence of new lesions (NLs) or progression of Non-target lesions (NTLs)
Time To Progress (TTP) | approximately 18 months
  TTP is defined as the time from randomization until the date of first documented disease progression (excluding death)
Overall Survival (OS) | From the date of first dose until the date of death from any cause or loss to follow-up, whichever comes first, assessed up to 100 months
  OS is defined as the time from randomization until death from any cause
Assessment of health-related quality of life (FACT-L) | approximately 18 months
  Change in FACT-L scores relative to Baseline
Safety variables | Assessments performed throughout the study period
  Adverse events, clinical symptoms, vital signs, ECG's, clinical laboratory safety tests, ect.
Plasma Concentrations of TY-9591 | approximately 18 months
  To characterise the pharmacokinetics (PK) of TY-9591
Plasma Concentrations of TY-9591-D1 | approximately 18 months
  To characterise the pharmacokinetics (PK) of TY-9591 metabolite D1
Plasma Concentrations of TY-9591-D2 | approximately 18 months
  To characterise the pharmacokinetics (PK) of TY-9591 metabolite D2

CONTACTS AND LOCATIONS:
Overall Officials: Baohui Han, MD, Principal Investigator — Shanghai Chest Hospital; Lin Wu, MD, Principal Investigator — Hunan Cancer Hospital
Locations (2):
- China (2):
  - Hunan Provincial Tumor Hospital, Changsha, Hunan
  - Shanghai Chest Hospital, Shanghai, Shanghai Municipality